CLINICAL TRIAL: NCT00003960
Title: Matched Unrelated and Haploidentical Bone Marrow Transplantation for Hematologic Malignancies
Brief Title: Donor Bone Marrow Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: J9828 CDR0000067159; P30CA006973 (NIH); JHOC-98032006; JHOC-J9828; NCI-G99-1543
Record Dates: First submitted 1999-11-01; First posted 2004-04-28 (Estimated); Last update posted 2014-05-02 (Estimated); Status verified 2014-05

CONDITIONS: Leukemia; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes
Keywords: refractory multiple myeloma; chronic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; acute undifferentiated leukemia; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Leukemia, Myeloid, Chronic-Phase; Anemia, Refractory, with Excess of Blasts; Leukemia, Biphenotypic, Acute | interventions — Busulfan; Cyclophosphamide; Methylprednisolone

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: methylprednisolone
Procedure: allogeneic bone marrow transplantation
Procedure: in vitro-treated bone marrow transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus donor bone marrow transplantation in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the 1-year survival rate of patients with hematologic malignancies after treatment with HLA-matched allogeneic bone marrow transplantation after high-dose chemotherapy.

OUTLINE: Patients receive oral busulfan four times a day on days -8 to -5, cyclophosphamide IV over 1 hour on days -4 to -1, and methylprednisolone IV over 1 hour every 12 hours on days -2 to 0. CD34+ stem cell augmented donor bone marrow is infused on day 0. Methylprednisolone is administered IV over 1 hour on days 5-16, and then tapered. Patients are followed every 6 months for 1 year and then annually thereafter.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of any of the following: Chronic myelogenous leukemia (CML) in first chronic phase Myelodysplastic syndrome Refractory anemia with excess blasts (RAEB) RAEB in transformation Secondary leukemias untreated or in complete remission 1 (CR1) Acute myeloid leukemia in complete remission 2 (CR2) Acute lymphocytic leukemia (ALL) in CR2 High-risk acute leukemia in CR1 Ph+ ALL in CR1 or consolidation after induction chemotherapy Must qualify for allogeneic bone marrow transplantation (BMT) No HLA-matched, sibling donor for BMT available No current CNS disease No history of more than 2 episodes of active CNS disease

PATIENT CHARACTERISTICS: Age: 19 to 55 Performance status: ECOG 0 or 1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin no greater than 2 mg/dL Renal: Creatinine no greater than 2 mg/dL Cardiovascular: LVEF at least 45% No active congestive heart failure, arrhythmia, or angina pectoris No myocardial infarction within the past 12 months Pulmonary: FEV1 and FVC at least 50% predicted (75% predicted if received prior thoracic or mantle radiotherapy) Other: No active serious infection (e.g., mucormycosis, uncontrolled aspergillosis, or tuberculosis) HIV negative Not pregnant Fertile patients must use effective contraception No concurrent debilitating medical or psychiatric illness that would preclude compliance No prior malignancy except curatively treated skin cancer or carcinoma of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No prior autologous or allogeneic bone marrow transplantation No prior transfusions from donor Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 1998-04; Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul V. O'Donnell, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Center for Cancer Treatment and Research, Columbia, South Carolina